CLINICAL TRIAL: NCT00109681
Title: A Randomized, Double-blind, Placebo-Controlled Phase II Study to Evaluate the Safety and Pilot Efficacy of Iloprost Inhalation Solution in Adults With Abnormal Pulmonary Arterial Pressure and Exercise Limitation Associated With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Inhaled Iloprost in Adults With Abnormal Pulmonary Pressure and Associated With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actelion (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ACTIVE C200-003
Record Dates: First submitted 2005-05-02; First posted 2005-05-03 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Pulmonary Fibrosis; Pulmonary Hypertension
Keywords: ACTIVE; iloprost; idiopathic pulmonary fibrosis; pulmonary arterial hypertension
MeSH Terms: conditions — Pulmonary Fibrosis; Hypertension, Pulmonary; Motor Activity; Idiopathic Pulmonary Fibrosis; Pulmonary Arterial Hypertension | interventions — Iloprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Iloprost Inhalation Solution (Ventavis)

SUMMARY:
The primary purpose of this study is to determine whether iloprost inhalation solution is safe in subjects with idiopathic pulmonary fibrosis (IPF) and elevated pulmonary arterial pressure. The secondary purpose is to evaluate the effectiveness of this treatment in subjects with this disease.

DETAILED DESCRIPTION:
While there are no FDA approved therapies for the treatment of IPF, there are therapies that have been shown to be effective in ameliorating the effects of pulmonary hypertension in patients with PAH (pulmonary arterial hypertension), including inhaled iloprost. However, these therapies have not been used extensively in patients with IPF who have pulmonary hypertension as a complication. The potential benefits of treatment of pulmonary hypertension complicating IPF include: improvement in pulmonary hemodynamics, with reduction in pulmonary artery pressure and pulmonary vascular resistance, and increase in cardiac output.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic pulmonary fibrosis according to American Thoracic Society criteria
* Diagnosis of elevated pulmonary pressures
* Six minute walk distance between 50-380
* NYHA functional class II - IV

Exclusion Criteria:

* Pulmonary fibrosis related to a systemic disorder
* Significant chronic obstructive pulmonary disease
* History of thromboembolic disease within the previous year
* Awaiting lung transplantation within next 36 weeks
* Active lung infection
* Survival prognosis of less than 1 year
* Significant left-sided heart failure, active coronary artery disease
* Clinically relevant liver disease
* Concurrent medications: epoprostenol, treprostinil, bosentan, PDE-5 inhibitor, investigational agents

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-04; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Safety

SECONDARY OUTCOMES:
6 minute walk distance
exercise associated oxygen desaturation

CONTACTS AND LOCATIONS:
Overall Officials: James Pennington, MD, Study Director — CoTherix
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCLA School of Medicine, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - The University of Chicago, Chicago, Illinois
  - University of Iowa College of Medicine, Iowa City, Iowa
  - Tulane University, New Orleans, Louisiana
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Mount Sinai Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Center at Tyler, Tyler, Texas
  - Inova Research Center, Church Falls, Virginia